CLINICAL TRIAL: NCT06821373
Title: Developing and Evaluating a Low-intensity Secondary Theory-based Chatbot Intervention to Reduce Common Digital Addictions, Sedentary Behaviors and Mental Distress Among Adolescents: A Randomized Controlled Trial
Brief Title: Chatbot Intervention to Reduce Common Digital Addictions, Sedentary Behaviors and Mental Distress Among Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Xue YANG, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20210481
Record Dates: First submitted 2025-02-04; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Internet Gaming Disorder; Social Media Addiction
Keywords: Internet gaming disorder; Chatbot; Social media addiction; Stage of change; motivation enhancement; Low-intensity; Sedentary lifestyle; Adolescent mental health
MeSH Terms: conditions — Internet Addiction Disorder; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Sham Comparator): Participants will receive educational but not SoC and MI-based materials about excessive digital use, IGD, and SMA. Such psycho-educational interventions are widely used in behavioral/mental health promotion and have been demonstrated to be effective in increasing knowledge and awareness of behavioral and mental problems. Based on a comprehensive literature review and our previous psycho-educational programs for behavioral/mental health promotion, the research team will design the psycho-educational materials. Themes include definitions, factors, and health consequences of excessive digital use, IGD, and SMA, information on healthy lifestyles, self-regulation skills, and help-seeking resources.
  Interventions: Behavioral: Control
- Chatbot (Experimental): The intervention includes five modules based on the five stages of Stages of change. Chatbots will build up a rapport with the participants, monitor their stage with a few simple questions based on previous Stages of Change studies, and provide stage-tailored packages of response, advice, and feedback (one of the five modules) accordingly to enhance their motivation and self-efficacy each week. For those who click 'yes' to a question assessing the first stage of change (PC), Chatbot will make a record and automatically ask questions assessing the next stage; for those who click 'no', Chatbot will automatically send them the module corresponding to their SoC via WhatsApp. Each module will take 10-15 minutes. In total, it will take 1 hour to complete all the modules.
  Interventions: Behavioral: Chatbot

INTERVENTIONS:
Behavioral: Chatbot — The intervention includes five modules based on the five stages of Stages of change. Chatbots will build up a rapport with the participants, monitor their stage with a few simple questions based on previous Stages of Change studies, and provide stage-tailored packages of response, advice, and feedback (one of the five modules) accordingly to enhance their motivation and self-efficacy each week. For those who click 'yes' to a question assessing the first stage of change (PC), Chatbot will make a record and automatically ask questions assessing the next stage; for those who click 'no', Chatbot will automatically send them the module corresponding to their SoC via WhatsApp. Each module will take 10-15 minutes. In total, it will take 1 hour to complete all the modules.
  Arms: Chatbot
Behavioral: Control — The intervention includes five modules based on the five stages of Stages of change. Chatbots will build up a rapport with the participants, monitor their stage with a few simple questions based on previous Stages of Change studies, and provide stage-tailored packages of response, advice, and feedback (one of the five modules) accordingly to enhance their motivation and self-efficacy each week. For those who click 'yes' to a question assessing the first stage of change (PC), Chatbot will make a record and automatically ask questions assessing the next stage; for those who click 'no', Chatbot will automatically send them the module corresponding to their SoC via WhatsApp. Each module will take 10-15 minutes. In total, it will take 1 hour to complete all the modules.
  Arms: Control

SUMMARY:
The goal of the study is to investigate the efficacy of a secondary low-intensity stage of change (SoC) and motivational interviewing (MI)-based Chatbot-assisted intervention in reducing digital addictions in adolescents with Internet gaming disorder (IGD) and/or social media addiction (SMA) by conducting a RCT.

Hypothesis: The intervention group will show a greater reduction in rates of IGD and/or SMA at post-treatment and 3-month follow-up than the control group.

Design and subjects: A two-armed RCT between the intervention group and psycho-educational control group for adolescents aged 10-19 with excessive screen time. Screening, baseline, post-programme, and 3-month follow-up evaluations will be conducted.

Participants will:

Be randomly assigned to online brief intervention or psycho-educational control

Complete questionnaires evaluating 1 ) Primary outcomes (IGD, SMA), 2) Secondary outcomes (sedentary lifestyle, mental distress, quality of life, eHealth literacy) and 3) Mediators/mechanisms (autonomy, competence)

ELIGIBILITY:
Inclusion Criteria:

* Students at grades 5-6 in primary schools or grades 7-12 in secondary schools,
* Positive screening results of IGD and/or SMA) based on the validated screening tools
* Using smartphone or Internet on a daily base, 4) students' and parental consent,
* Chinese speaking.

Exclusion Criteria:

* Current use of any psychotropic medication.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Internet gaming disorder (IGD) | From enrollment to the end of follow-up at 3 months
  IGD symptoms are assessed using the Nine-Item Internet Gaming Disorder Scale-Short Form (IGDS9-SF) consists of nine questions that assess IGD symptoms, including preoccupation, tolerance, withdrawal, unsuccessful attempts to limit gaming, deception or lies about gaming, loss of interest in other activities, use despite knowledge of harm, use for escape or relief of negative mood, and harm. The response options for each item include "yes=1" and "no=0". The overall score of the scale ranges from 0 to 9, with a higher score implying a higher level of IGD symptoms. Participants with score ≥ 5 will be classified as having probable IGD.
Social media addiction (SMA) | From enrollment to end of follow-up at 3 months
  SMA is defined as excessive use of social media with the addictive symptoms like mood modification, salience, tolerance, withdrawal symptoms, conflict, and relapse. The symptoms of SMA will be measured by the 6-item Bergen Social Media Addiction Scale (BSMAS) based on the six core components of addictive behaviors, including cognitive salience, tolerance, mood modification, difficulty in regulating use, withdrawal, and interference with role performance. The items are rated using a Likert type scale ranging between 1 (very rarely) and 5 (very often). A higher sum score in the BSMAS indicates a greater likelihood of being at risk of developing social media addiction. A cut-off score over 19 indicates probable SMA.
Composite score of IGD and SMA | From enrollment to end of follow-up at 3 months.
  Composite outcome of IGD score and SMA score: we define a simple composite as the sum of the two outcomes. Because each outcome measure uses a different scale and has different statistical properties, we will standardize the two variables (i.e., scores of IGD and SMA) first, and then combine the two standardized scores of the outcomes into a composite.

SECONDARY OUTCOMES:
Sedentary lifestyle | From enrollment to end of 3 months follow-up
  Sedentary behavior is defined as any waking behavior such as sitting or leaning with an energy expenditure of 1.5 metabolic equivalent task (MET) or less. Sedentary lifestyles will be measured by the 10-item sedentary lifestyles questionnaire (SLQ) which has been used in Chinese school children. Subjects will report the average daily time spent (hours) during the weekdays and weekends in the following activities: Using smartphone or tablet PC for learning/doing paper homework or reading or writing/ sedentary leisure time without time for screen leisure. Average number of daily hours will be calculated as (total sedentary weekday hours × 5 + total sedentary weekend hours × 2) ÷ 7.
Entertainment screen time | From enrollment to end of follow-up at 3 months
  The American Academy of Pediatrics has recommended that time allotted to Internet gaming or the total amount of entertainment screen time in general (e.g., using social media platforms/social networking sites, watching TV/videos) should be <1 to 2 hours per day for children and adolescents given the significant health consequences of excessive Internet gaming and screen time. Thus, participants who report the total amount of entertainment screen time with two or more hours per day will be classified as excessive screen time cases and positive cases in our school-based screening.
Health-related Quality of life | From enrollment to end of follow-up at 3 months
  Quality of life will be measured by the EQ-5D-Y scale (Y for youth). The EQ-5D-Y uses a similar 5-dimenional descriptive system with the EQ-5D but child-friendly wording, referring to mobility ('walking about'), self-care ('looking after myself'), usual activities ('doing usual activities'), pain and discomfort ('having pain or discomfort'), and anxiety and depression ('feeling worried, sad or unhappy'). Each dimension includes one item which has three functioning levels: no problem, some problems, and a lot of problems. The EQ-5D-Y also includes an easily understandable modification of the vertical, graduated Visual Analogue Scale (VAS) of EQ-5D, where the respondent rates his or her overall health status on a scale from 0 to 100 with 0 representing the worst and 100 the best health state the individual can imagine.
Mental distress | From enrollment to end of follow-up at 3 months
  Mental distress is defined as a collection of mental problems that may not fall into standard diagnostic criteria and are characterized by symptoms of sleeplessness, depression, anxiety, exhaustion, irritability, poor memory, difficulty in concentrating, and somatic complaints. The Chinese K6 questionnaire comprises six questions that ask respondents to rate how frequently they have felt 'nervous', 'hopeless', 'restless or fidgety', 'so depressed that nothing could cheer you up', 'that everything was an effort', and 'worthless' during the past 30 days. Response options included 'none of the time' (0), 'a little of the time' (1), 'some of the time' (2), 'most of the time' (3), and 'all of the time' (4). The range of score for K6 was thus from 0 to 24.
eHealth literacy | From enrollment to end of follow-up at 3 months
  eHealth literacy is defined as the ability of individuals to seek, find, understand, and appraise health information from electronic sources and apply such information to addressing or solving a health problem. eHealth literacy will be assessed by the 8-item eHealth Literacy Scale (eHEAL), which was validated in Chinese student population. The sample items include 'I know how to find helpful resources on the internet' and 'I know how to use the internet to answer my questions about health'. Ratings were made on 5-point Likert scales, ranging from 1= strongly disagree to 5 = strongly agree, with higher scores indicating a higher level of eHealth literacy.

OTHER OUTCOMES:
Autonomy | From enrollment to end of follow-up at 3 months
  Autonomy involves feeling a sense of personal agency and volition such that one's behavior is perceived to emanate from an internal locus of causality. To assess autonomy to reduce dependence on Internet gaming/social media, the subscale of the Psychological Need Satisfaction in Exercise Questionnaire (PNS-A) will be adapted and used. The Chinese version was demonstrated to have good psychometric properties. The scale includes six items measuring psychological need fulfillment of autonomy. Items are rated on a 6-point Likert scale, ranging from 1 (false) to 6 (true). Total scores range from 6 to 36, with higher scores being indicative of higher degrees of autonomy.
Competence (self-efficacy) | From enrollment to end of follow-up at 3 months
  Competence refers to interacting effectively with one's environment while mastering challenging tasks. The 6-item competence subscale of PNS (PNS-C) will be used to assess competence to reduce dependence on Internet gaming/social media. Total scores range from 6 to 36, with higher scores being indicative of higher degrees of autonomy or competence.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Yang, Doctoral, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- JC School of Public Health and Primary Care, The Chinese University of Hong Kong, Hong Kong, Hong Kong